CLINICAL TRIAL: NCT06166303
Title: Effect of Number of Previous Cesarean Sections on the Results of Angiogenic Factors. A Descriptive, Prospective Study.
Brief Title: Number of Previous Cesarean Sections on the Results of Angiogenic Factors.
Status: Not yet recruiting | Type: Observational
Sponsor: Saint Thomas Hospital, Panama (Other)
Responsible Party: Principal Investigator, Osvaldo A. Reyes T., Head of the research deparment, Saint Thomas Hospital, Panama
Other Study IDs: U1111-1301-2580
Record Dates: First submitted 2023-12-04; First posted 2023-12-12 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Cesarean Section
Keywords: Cesarean section; Angiogenic factors; Preeclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Previous Cesarean Section: Subjects with one or more previous cesarean sections
  Interventions: Diagnostic Test: sFlt-1/PGIF
- No Cesarean: Subjects scheduled for an elective or urgent cesarean, but no history of previous cesarean section
  Interventions: Diagnostic Test: sFlt-1/PGIF

INTERVENTIONS:
Diagnostic Test: sFlt-1/PGIF — Index of sFlt-1/PGIF

SUMMARY:
Hypertensive disorders of pregnancy (HPT) are an important cause of maternal-feto-neonatal morbidity and mortality, being one of the three leading causes of maternal death in our country and in developing countries. The only cure for THE is termination of pregnancy, which ends up being a decision in which gestational age and maternal risks must be balanced. Angiogenic factors have come to occupy an indispensable place in the arsenal of tools that can be used to separate the patient with a high likelihood of complications from those in whom prolongation of pregnancy could represent an important neonatal benefit.

Although the usefulness of angiogenic factors in these scenarios is known, little is known about the effects that other conditions might have on their serum levels, mainly those that have an effect on trophoblastic invasion, the process that initiates implantation of the pregnancy in the endometrium. The purpose of the present study is to assess the effect that a history of uterine surgery, such as caesarean section, might have on angiogenic factor scores in subjects with no history of a hypertensive disorder of pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* 36 weeks of gestation or more
* Singleton pregnancy
* Previous cesarean section (case)

Exclusion Criteria:

* Vasculitis
* Twin pregnancy
* Chronic endometritis
* Smoking
* Lupus
* Renal failure
* Liver disease
* Thrombocytopenia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant woman with a previous cesarean section
Sampling Method: Probability Sample
Enrollment: 540 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Index sFlt-1/PIGF | From the moment of randomization up until delivery. Between 24-48 hours.
  Angiogenic factors, normal value.

SECONDARY OUTCOMES:
Progression to preeclampsia | Up until discharge. On average, 7 days
  Number of subjects that develop a preeclampsia

CONTACTS AND LOCATIONS:
Overall Officials: Osvaldo Reyes, Principal Investigator — Hospital Santo Tomás
Locations (1):
- Saint Thomas H, Panama City, Provincia de Panamá, Panama

IPD SHARING:
Plan to Share IPD: No